CLINICAL TRIAL: NCT03677037
Title: Short-term Versus Long-term Mentalization-based Therapy for Outpatients With Subthreshold or Diagnosed Borderline Personality Disorder: a Randomized Clinical Trial
Brief Title: The Short-Term MBT Project
Acronym: MBT-RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: University of Copenhagen (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-18023136
Record Dates: First submitted 2018-09-14; First posted 2018-09-19 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Borderline Personality Disorder
Keywords: mentalization-based therapy; borderline personality disorder; randomized clinical trial; psychotherapy research; treatment intensity
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-term MBT (Experimental): The experimental group is short-term mentalization-based therapy. The treatment program includes 20 weeks of mentalization-based group therapy with conjoined individual therapy every second week. The program also includes psychoeducation and individual caseformulations.
  Interventions: Other: Short-term MBT
- Long-term MBT (Active Comparator): The control group is long-term mentalization-based therapy. The treatment program includes 14 months of weekly mentalization-based group therapy with combined individual therapy every second week. The program also includes psychoeducation and individual caseformulations.
  Interventions: Other: Long-term MBT

INTERVENTIONS:
Other: Short-term MBT — Short-term mentalization-based therapy
  Arms: Short-term MBT
Other: Long-term MBT — Long-term mentalization-based therapy
  Arms: Long-term MBT

SUMMARY:
The study will evaluate the benefitial and harmful effects of short-term (20 weeks) compared to long-term (14 months) mentalization-based therapy for outpatients with subthreshold or diagnosed borderline personality disorder.

DETAILED DESCRIPTION:
Psychotherapy for borderline personality disorder is often lengthy and resource-intensive. Mentalization-based therapy is an example of an evidence-based treatment that currently has empirical support as an 18-months outpatient program for borderline personality disorder. However, this duration is rarely available, and the long and costly treatment combined with a highly prevalent disorder result in insufficient access to evidence-based care.

The trial is an investigator-initiated, single-centre, assessor-blinded, randomized clinical superiority trial of short-term (20 weeks) compared to long-term (14 months) outpatient mentalization-based therapy for borderline personality disorder or subthreshold borderline personality disorder. Participants will be recruited from the Outpatient Clinic for Personality Disorders at Stolpegaard Psychotherapy Centre, Mental Health Services, Capital Region of Denmark. Participants will be assessed at trial intake using the Mini International Neuropsychiatric Interview and the Structured Clinical Interview for DSM-5 Personality Disorders. Participants will be included if they meet a minimum of four DSM-5 criteria for borderline personality disorder. Participants will be assessed blind to treatment allocation at baseline, and at 8, 16, and 24 months after randomization.

The primary outcome is severity of borderline symptomatology assessed using the Zanarini Rating Scale for Borderline Personality Disorder interview. Secondary outcomes include self-harm incidents, functional impairment (Work and Social Adjustment Scale), quality of life (Short-Form Health Survey), and global functioning (Global Assessment of Functioning scale). Psychiatric symptoms (Symptom Checklist 90) will be included as an exploratory outcome. Measures of personality functioning, attachment, group alliance, borderline symptoms and mentalization skills will be included as predictor and mediator variables.

ELIGIBILITY:
Inclusion Criteria exclusive to the Outpatient Clinic

* Age >18 years
* Personality disorder(s) considered to be primary diagnosis/diagnoses

Inclusion Criteria exclusive to the trial:

* A minimum of four DSM-5 criteria for borderline personality disorder
* Written informed consent

Exclusion Criteria exclusive to the Outpatient Clinic:

* Possibility of a learning disability (IQ<75)
* A diagnosis of schizotypal personality disorder or antisocial personality disorder
* Presence of a comorbid psychiatric disorder that requires specialist treatment elsewhere
* Current (past 2 months) substance dependance including alcohol
* Concurrent psychotherapeutic treatment outside the clinic

Exclusion Criteria exclusive to the trial:

- Lack of informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in severity of borderline personality disorder assessed with the Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) interview | Assessed at baseline, and at 8, 16 and 24 months post-randomization
  ZAN-BPD is an investigator-administered interview assessing change in severity of borderline personality disorder over time. Each of the nine DSM-5 criteria for borderline personality disorder are rated on a scale from 0-4, where 4 is the most severe, yielding a total score from 0-36.

SECONDARY OUTCOMES:
Change in functional impairmment assessed with the Work and Social Adjustment Scale (WSAS) | Assessed at baseline, and at 8, 16 and 24 months post-randomization
  WSAS is a 5-item questionnaire assessing change in functional impairment. Each item is rated on a scale from 0-8, where 0 is no impairment and 8 is severe impairment, yielding a total score between 0-40.
Change in quality of life assessed with the Short-Form Health Survey 36 (SF-36) | Assessed at baseline, and at 8, 16 and 24 months post-randomization
  SF-36 is a questionnaire assessing change in self-reported quality of life over time. The instrument measures eight health dimensions: physical function (PF), role physical (RF), bodily pain (BP), social function (SF) role emotional (RE), general health (GH), vitality (VT) and mental health (MH). The questions related to each dimension are scored on a scale from 0 (worst score) to 100 (best score).
Change in global functioning assessed with the Global Assessment of Functioning (GAF) | Assessed at baseline, and at 8, 16 and 24 months post-randomization
  GAF is an investigator-administered rating of change in global functioning over time. Global funtioning is rated on a scale from 0-100 for both symptomatic and functional impairment, yielding two total scores from 0-100, where 100 is no impaitment and 0 is severe impairment.
Change in amount of self-harm incidents | Assessed at baseline, and at 8, 16 and 24 months post-randomization
  Proportion of participants with severe self-harm defined as deliberate acts of self-harm resulting in visible tissue damage - data will be collected as both dichotomous data and count data.

OTHER OUTCOMES:
Change in psychiatric symptom distress assessed with the Symptom Checklist 90 (SCL-90) | Assessed at baseline, and at 8, 16 and 24 months post-randomization
  SCL-90 is a questionnaire assessing change in psychiatric symptom distress over time. All 90 items are rated on a scale from 0-4. The total score is divided by number of items, yielding a total score on the Global Severity Index ranging from 0 to 4, where 4 is the most severe.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Simonsen, PhD, Study Director — Sponsor-Investigator
Locations (1):
- Stolpegaard Psychotherapy Centre, Mental Health Services, Capital Region of Denmark, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Juul S, Jakobsen JC, Hestbaek E, Jorgensen CK, Olsen MH, Rishede M, Frandsen FW, Bo S, Lunn S, Poulsen S, Sorensen P, Bateman A, Simonsen S. Short-Term versus Long-Term Mentalization-Based Therapy for Borderline Personality Disorder: A Randomized Clinical Trial (MBT-RCT). Psychother Psychosom. 2023;92(5):329-339. doi: 10.1159/000534289. Epub 2023 Nov 7. PMID 37935133
- [Derived] Juul S, Simonsen S, Poulsen S, Lunn S, Sorensen P, Bateman A, Jakobsen JC. Detailed statistical analysis plan for the short-term versus long-term mentalisation-based therapy for outpatients with subthreshold or diagnosed borderline personality disorder randomised clinical trial (MBT-RCT). Trials. 2021 Jul 28;22(1):497. doi: 10.1186/s13063-021-05450-y. PMID 34321051
- [Derived] Gibbon S, Khalifa NR, Cheung NH, Vollm BA, McCarthy L. Psychological interventions for antisocial personality disorder. Cochrane Database Syst Rev. 2020 Sep 3;9(9):CD007668. doi: 10.1002/14651858.CD007668.pub3. PMID 32880104
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Juul S, Lunn S, Poulsen S, Sorensen P, Salimi M, Jakobsen JC, Bateman A, Simonsen S. Short-term versus long-term mentalization-based therapy for outpatients with subthreshold or diagnosed borderline personality disorder: a protocol for a randomized clinical trial. Trials. 2019 Apr 5;20(1):196. doi: 10.1186/s13063-019-3306-7. PMID 30953536